CLINICAL TRIAL: NCT03876795
Title: Evaluation of Effectiveness of Combined Intra-articular and Intra-osseus Injection VS a Single Intra-articular Injection of Bone Marrow Concentrate for the Treatment of Osteoarthritis in the Knee. (INTERFACE) Double Blind, Randomized Clinical Trial
Brief Title: Evaluation of Effectiveness of Combined Intra-articular and Intra-osseus Injection VS a Single Intra-articular Injection of Bone Marrow Concentrate
Acronym: INTERFACE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INTERFACE
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Osteoarthritis, Knee
Keywords: Bone Marrow Comcentrate; intra-articular; intra-osseus
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single intra-articular Bone Marrow Concentrate injection (Active Comparator): Single intra-articular Bone Marrow Concentrate injection in the knee
  Interventions: Biological: Bone Marrow Concentrate
- combined Bone Marrow Concentrate injection (Experimental): combined Bone Marrow Concentrate injection (intra-articular and intra-osseus)
  Interventions: Biological: Bone Marrow Concentrate

INTERVENTIONS:
Biological: Bone Marrow Concentrate — Bone Marrow Concentrate injection

SUMMARY:
Osteoarthritis (OA) is one of the most common diseases resulting in large burdens on society.

Among the emerging treatments, Bone Marrow Concentrate (BMC) intra-articular injections are a promising regenerative approach. However, they offer only a temporary benefit since they target synovial and chondral tissues but fail to address the osteochondral interface, which plays a key role in the onset and progression of joint degeneration.

This project will investigate the efficacy of combined BMC injections, targeting both intra-articular tissues and subchondral bone, to treat OA in a Randomized Controlled Trial (RCT).

DETAILED DESCRIPTION:
The main aim is to evaluate in a RCT the potential of a new combined BMC treatment for OA, through the use of scores for the clinical outcome, the study of imaging and biological samples for tissue regeneration and systemic effects, and the identification of BMC and patient characteristics predictive of better results.

All patients will undergo an arthroscopic procedure to debride degenerated tissues (this can offer a temporary benefit but not long lasting results) before BMC intra-articular injection. Half patients will receive also the injection of BMC at the subchondral level (bone samples obtained to allow BMC placement will be sent to the Lab).

The same minimally invasive incisions will be used for all patients, ensuring patient blinding. Evaluations, performed by medical staff not involved in the treatment to ensure double blinding, will document subjective clinical improvement, functional measurements, biomarker study, and imaging with the use of modern 3TMRI and qCT technology. BMC characterization and patient features will be analysed to identify factors predictive of a better outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, aged between 40 and 70;
2. Arthrosis of the medial compartment (grade 2-3 according to the Kellgren-Lawrence score> 4 months);
3. Failure after at least 6 months of conservative treatment (drug therapy with NSAIDs and painkillers, hyaluronic acid infiltration, corticosteroid infiltration, PRP);
4. Patients' ability and consent to participate in clinical and radiological follow-up;
5. Signature of informed consent.

Exclusion Criteria:

1. Patients with trauma in the 6 months prior to surgery;
2. Patients with maligncy;
3. Patients suffering from rheumatic diseases;
4. Patients suffering from non-compensated diabetes;
5. Patients suffering from uncompensated thyroid metabolic disorders;
6. Patients abusing alcoholic beverages, drugs or drugs;
7. Patients with axial deviations> 5 °;
8. Body Mass Index> 35;
9. Patients treated with joint infiltrations in the previous 6 months;
10. Patients treated with surgery at the same knee in the previous 12 months.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
change of Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score trend over time | basal 2,6,12 months after treatment
  WOMAC is a validated score, designed to highlight the problems of patients with lower limb pathologies, in particular in terms of pain, stiffness and functionality. The score will be completed by the patient, possibly in the presence of an investigator, and simple guidelines for self-compilation will be provided.

SECONDARY OUTCOMES:
IKDC Subjective Knee Evaluation Form (IKDC) | 2,6,12 months
  IKDC is a validated score used in the evaluation of symptoms, function and sport activity in patients suffering of knee diseases, such as meniscal or ligamentous damage, osteoarthritis. The Subjective Knee Form provides the best method of overall assessment of the most significant symptoms and disabilities for a population that has undergone cartilage repair treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- Rizzoli Orthopaedic Institute, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silva S, Andriolo L, Boffa A, Di Martino A, Reale D, Vara G, Miceli M, Cavallo C, Grigolo B, Zaffagnini S, Filardo G. Prospective double-blind randomised controlled trial protocol comparing bone marrow aspirate concentrate intra-articular injection combined with subchondral injection versus intra-articular injection alone for the treatment of symptomatic knee osteoarthritis. BMJ Open. 2022 Sep 8;12(9):e062632. doi: 10.1136/bmjopen-2022-062632. PMID 36468635